CLINICAL TRIAL: NCT02516059
Title: Does Postoperative Administration of Oral Oxycodone With/Without Naloxone, Reduce the Duration of Epidural Analgesia in Patients Undergoing Cystectomy Without Impairing Its Benefits? A Randomized, Double Blind Controlled Trial
Brief Title: Early Postoperative Administration of Oxycodone +/- Naloxone and Duration of Epidural Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 068/15; WUPD 01-14 (Other: Inselspital); 2015DR4112 (Other: Swissmedic)
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Postoperative Pain Management; Radical Cystectomy; Epidural Analgesia; Oral Oxycodone With/Without Naloxone; Return of the Bowel Function
Keywords: thoracic epidural analgesia; oxycodone; oral naloxone; radical cystectomy; bowel function; pain
MeSH Terms: conditions — Pain | interventions — Oxycodone; Naloxone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxycodone and naloxone (Targin®) (Active Comparator): Oxycodone and naloxone (Targin®; Mundipharma Medical Company and Mundipharma Research GmbH & Co Basel, Switzerland): Will be orally administered at 12 hours intervals, starting with 10mg/5mg on POD 3 and move to 20mg/10mg the other day.
  Interventions: Drug: oxycodone/naloxone; Device: epidural catheter
- Oxycodone (Oxycontin®) (Active Comparator): Oxycodone (Oxycontin®, Mundipharma Medical Company and Mundipharma Research GmbH & Co Basel, Switzerland): Will be orally administered at 12 hours intervals, starting with 10 mg on POD 3 and move to 20 mg the other day.
  Interventions: Drug: Oxycodone; Device: epidural catheter
- Placebo (Placebo Comparator): Placebo (Mundipharma Medical Company and Mundipharma Research GmbH & Co Basel, Switzerland): Will be orally administered at 12 hours intervals starting on POD 3.
  Interventions: Drug: Placebo; Device: epidural catheter

INTERVENTIONS:
Drug: oxycodone/naloxone — Oxycodone and naloxone (Targin®; Mundipharma Medical Company and Mundipharma Research GmbH & Co Basel, Switzerland): Will be orally administered at 12 hours intervals, starting with 10mg/5mg on POD 3 and move to 20mg/10mg the other day.
  Other Names: Targin®
  Arms: Oxycodone and naloxone (Targin®)
Drug: Oxycodone — Oxycodone (Oxycontin®, Mundipharma Medical Company and Mundipharma Research GmbH & Co Basel, Switzerland): Will be orally administered at 12 hours intervals, starting with 10 mg on POD 3 and move to 20 mg the other day.
  Other Names: Oxycontin®
  Arms: Oxycodone (Oxycontin®)
Drug: Placebo — Placebo (Mundipharma Medical Company and Mundipharma Research GmbH & Co Basel, Switzerland): Will be orally administered at 12 hours intervals starting on POD 3.
  Arms: Placebo
Device: epidural catheter

SUMMARY:
Cystectomy with urinary diversion (ileal conduit, ileal orthotopic neobladder, catheterizable ileal pouch) is major abdominal surgery, which is associated with a high incidence of gastrointestinal complications.Perioperative techniques aiming at an early return of bowel function are to be pursued.

Optimal postoperative pain management is one of the key factors leading to enhanced recovery after surgery. The perioperative use of an epidural analgesia for major abdominal surgery is established, not only because of its excellent analgesic properties, but also because it can accelerate the return of bowel function. However, epidural analgesia is associated with additional costs, need for close monitoring and nursing. In addition each supplemental day with an indwelling epidural catheter increases the risk of infection. So it is recommended to re-assess the risk/benefit ratio of an epidural analgesia after 4 days, if not sooner. Therefore, it is important to develop strategies that reduce its duration without impairing the benefits. Systemic analgesics with prolonged-release oral formulation like oral oxycodone (Oxycontin®) or combined drug mixture (oral oxycodone/naloxone (Targin®)) could be a valuable alternative pain treatment as a second analgesic step, starting on postoperative day (POD) 3, so that the epidural catheter could be removed earlier without impairing postoperative enhanced recovery including return of the bowel function. Both oxycodone and naloxone orally administered are a recognized and accepted treatment option.

The objective of this study is to evaluate the implementation of an oral opioid with or without naloxone in the early postoperative period in patients undergoing open radical cystectomy with urinary diversion and intraoperative and early postoperative use of epidural analgesia. The investigators expect an unchanged early return of the bowel function and equal analgesia with a reduced length of stay of the epidural catheter (primary endpoint), thus potentially reducing epidural catheter associated complications and lowering costs (nursing and pain service).

DETAILED DESCRIPTION:
Background

Cystectomy with pelvic lymph node dissection and urinary diversion is major abdominal surgery, which is associated with a high incidence of postoperative complications. Gastrointestinal complications are frequent and perioperative techniques aiming at an early return of bowel function are to be pursued.The rationale for this patients population (i.e. cystectomy patient with ileal urinary derivation) is that they are at high risk for postoperative complications (around 50%) and specially gastrointestinal (8-20%). There is a need for improvement in the postoperative setting aiming to reduce complications and costs.

Optimal postoperative pain management is one of the key factors leading to enhanced recovery after surgery. The perioperative use of thoracic epidural analgesia (TEA) for major abdominal surgery is established, not only because of its excellent analgesic properties, but also because TEA reduces the postoperative stress response, accelerates the return of bowel function, and lowers postoperative morbidity and mortality. However, TEA is associated with additional costs, need for close monitoring and nursing. Once successfully established, TEA requires constant attention from skilled nurses and anaesthetists often from an acute pain service to achieve and maintain optimal analgesia. Attention must also be directed to limiting or avoiding side-effects such as hypotension or motor block, which will reduce the benefits of the technique by preventing the patient from mobilizing effectively after operation.In addition each supplemental day with an indwelling TEA catheter increases the risk of infection, which is associated with a high morbidity. The mean length of stay of the TEA catheter in cystectomy patients at the investigators' institution is 6 days. If the risk of epidural infection is low (estimated 1:2000 in Switzerland, this risk increases the longer the epidural catheter is left in place. It is recommended to re-assess the risk/benefit ratio of TEA after 4 days, if not sooner. Therefore, it is important to develop strategies that reduce the duration of TEA without impairing the benefits. Enhanced recovery after surgery protocols, which have been established for colorectal surgery in the last 10 years, recommend removing the TEA catheter in the morning of postoperative day (POD) 2, which does not impair the return of the gastrointestinal function. However, while this approach is well established for colorectal surgery, there is less evidence for small bowel surgery or cystectomy with urinary diversion.

Systemic analgesics with prolonged-release oral formulation like oral oxycodone (Oxycontin®) or combined drug mixture (oral oxycodone/naloxone (Targin®)) could be a valuable alternative pain treatment as a second analgesic step, starting on POD 3, so that the epidural catheter could be removed earlier without impairing postoperative enhanced recovery including return of the bowel function. Both oxycodone and naloxone orally administered are a recognized and accepted treatment option.The selected dosages of both orally administered drugs are in accordance with the literature and follow the recommendation of the manufacturers. In addition the dosages reflect the clinical practice of the investigators' institution. These drugs are daily used in a clinical setting in their pain service. The implementation of a placebo controlled group is considered as a gold standard approach in a randomized controlled trial aiming to assess the benefit of a drug for a specific indication. In addition, a rescue pain medication is implanted in the protocol. Rescue medication for breakthrough pain will be additional epidural boluses of 5 ml, limited to maximum one bolus per h. In case of persistent pain, orally administered of 5 mg oxycodone every 4-6 hours will be allowed by the ward nurses.

The investigators expect, by administering oxycodone/naloxone in the early postoperative period to reduce the length of TEA without impairing the return of the bowel function. This could reduce the risk induced by the prolonged TEA (i.e. local infection, malfunction) and costs (pain service). This can result in the implementation in the future of a new postoperative analgesia concept with the early postoperative administration of an oral pain killer, reducing the length of epidural analgesia without impairing the enhanced recovery.

A total of 90 patients (30 per group) undergoing cystectomy with urinary diversion with perioperative thoracic epidural analgesia will be studied.

Blinding:

Batches and blinding will be organized by Mundipharma Medical Company (Basel, Switzerland) and provided by Mundipharma Research GmbH & Co. KG granting good manufacturing practice (GMP). As Targin tablets are oblong in shape and the Oxycontin tablets are round a double dummy approach is inevitable to warrant the fully blinding. It will not be able to optically recognize the type of drugs administered. The one will contain only placebo, the second 20mg of oxycodone (Oxycontin®) and the third a mixture of oxycodone (20mg) and naloxone (10mg) (Targin®). Drugs will be orally administered at 12 hours intervals.

Study nurses on the Department of Urology will bring the randomized blinded drugs to the intermediate care unit in a sealed package, only described with only the name of the included patient.

This will allow for blinding of the patient, the patient's nurses of the IMC and ward and urologist, and data assessor (including pain service).

Randomisation will be done by computer generated list, with blocks of 10 patients; allocation will be left in concealed opaque and numbered envelopes. Patients will be included strictly according to the lowest number.

Duration of the study:

The annual case load of cystectomy is around 100 in the investigators' institution per year. The investigators expect to recruit the participants within 24 months. To ensure that the study can be conducted in the anticipated timeframe, an interim analysis of recruitment is scheduled 1 year after Swissmedic study approval. If the recruitment remains below expectations and completion of the study in a timely manner is jeopardized, this would result in abandoning the Oxycodone arm.

Sequence of the study:

Seven days (inclusion the day before surgery, finished after removal of the epidural catheter)

Time course of the study:

Admission day:

After informed patient consent, patients will be randomized.

End of surgery till POD 3, morning:

The study will start after cystectomy combined with urinary diversion is successfully performed in combined anesthesia (general plus TEA). After closure of the abdominal wall, continuous epidural analgesia will be maintained with bupivacaine 1.25mg/ml using an ambulatory infusion pump. The initial infusion rate will be 8 ml/h, with additional bolus volumes of 4 ml (lockout time: 1 h). The infusion rate can be adapted if necessary based on assessments made every 4 h to maintain a pain intensity lower than 3 at rest and lower than 5 during mobilization on the numeric rating scale (NRS), where 0=no pain and 10=worst pain imaginable. The maximum infusion rate will be 10 ml/h. This epidural treatment is in accordance with the investigators' internal standard and has been successfully implemented in the last 15 years. Data on pain intensity, amount of epidural mixture used per 24 h and use of rescue analgesics will be recorded daily. In addition, episodes of PONV, first flatus and defecation and body weight will be documented.

POD 3 around 08:00 a.m.:

According to the randomization, patients will receive blinded batches with 20mg oxycodone, 20mg oxycodone plus 10mg naloxone or oral placebo every 12 h, starting with 10 mg bid respectively 10mg/5mg and move to 20 mg bid (20mg/10mg) the other day. Epidural mixture infusion will be reduced in steps of 2 ml according to the NRS score to maintain a pain intensity lower than 3 at rest and lower than 5 during mobilization during 6 h. The epidural catheter will be removed when during 6 h the rate is 2 ml/h, and the patient has a NRS < 3 and < 5 at rest and during mobilisation, respectively. If the epidural catheter cannot be removed because of the subcutaneous administration of low weighted molecular heparin (LWMH) (always around 20:00), the infusion will be stopped (0 ml/h) and the length of stay of the epidural catheter registered (length of stay of the epidural catheter= insertion of the catheter to rate of epidural mixture =0ml/h), and the catheter will be removed according to the investigators' internal guideline (at least 12 h after subcutaneous administration of LWMH). The time the epidural infusion was stopped will be recorded as removal of the epidural catheter.

Objective

The objective of this study is to evaluate the implementation of an oral opioid with or without naloxone in the early postoperative period in patients undergoing cystectomy and urinary diversion with intraoperative and early postoperative use of TEA. The investigators expect an unchanged early return of the bowel function and equal analgesia with a reduced length of stay of the epidural catheter (primary endpoint), thus potentially reducing epidural catheter associated complications and lowering costs (nursing and pain service).

Methods

Trial design:

Randomized, double blind, parallel groups, single center, intervention placebo controlled study

Setting:

Single center: Department of Urology, University Hospital Bern, Inselspital.

Selection of the trial subjects:

A total of 90 patients (30 per group) undergoing cystectomy with urinary diversion with perioperative thoracic epidural analgesia will be studied.

Phase 4 For clinical trials with drugs: Clinical study phase or phase of clinical development (e.g. Phase 1, 2, 3 or 4; or according to ICH E8 para 3.1.3 Human Pharmacology, Therapeutic Exploratory, Therapeutic Confirmatory or Therapeutic Use); in case of Medical Device study rename and use e.g. "Phase of development".

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Informed Consent as documented by signature
* Renal function: eGFR >40ml/min
* Normal liver function
* Cystectomy with urinary diversion
* Use of thoracic epidural analgesia

Exclusion Criteria

* Contraindications to the class of drugs under study, e.g. known hypersensitivity or allergy to class of drugs or the investigational product, i.e. known allergy to oxycodone naloxone or other excipients
* Women who are pregnant or breast feeding, (exclusion for surgery per se)
* Known or suspected non-compliance, drug or alcohol abuse
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, severe psychiatric disorder, etc. of the participant
* Severe asthma bronchiale, severe COPD
* Severe respiratory depression with hypoxia and/or hypercapnoea, cor pulmonale
* Preoperative use of MAO-Inhibitors (or has to be stopped 2 weeks before surgery)
* Patients with chronic pain
* Patients with regular use of antiemetics, laxatives, opioids or other types of analgesics
* Preoperative regular use of non steroidal anti inflammatory drugs and steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2017-02-20 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Length of stay of the epidural catheter in days | At removal of the catheter, expected to be on average of 6 days

SECONDARY OUTCOMES:
Pain scores (NRS 0-10) at postoperative day (POD) 1 to POD 7 | From postoperative day (POD) 1 to 7
  Measured in numeric rating score NRS; measured by questionnaire
Duration of the return of the bowel function in days | From postoperative day (POD) 1 to 7

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y Wuethrich, MD, Principal Investigator — Department of Anaesthesiology and Pain Therapy, University Hospital Bern; Fiona C Burkhard, MD, Study Director — Department of Urology, University Hospital Bern
Locations (1):
- Dep of Urology Bern University Hospital, Bern, Switzerland